CLINICAL TRIAL: NCT01045512
Title: The Role of the "Inflammatory/ Pathogen Burden" for Cardiac Ageing
Acronym: AntiCardAgeing
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unsufficient recruitment
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KKSH-38; 2007-003003-12 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Aging; Inflammation
Keywords: immunosenescence; heart rate variability; autonomic nervous system; ageing; inflammatory/pathogen burden; physical activity
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- statins, standardised physical training (Active Comparator)
  Interventions: Drug: fluvastatin
- to continue with current lifestyle (No Intervention)

INTERVENTIONS:
Drug: fluvastatin — 40-80mg once daily
  Arms: statins, standardised physical training

SUMMARY:
In the elderly a chronic basal systemic inflammation prevails - which is evident by enhanced CRP or IL-6 plasma concentrations - and by compromised defense mechanisms against invading microbes. These alterations belong to the physiological ageing process of the immune system (immunosenescence) and are regarded as an inflammatory response towards lifelong antigen stress ("inflammatory/pathogen burden"). This lifelong antigen stress evokes an age-dependent basal inflammatory activation of innate immunity as well as a wasting of specific immunity: it is supposed that in the course of life-time due to a multitude of infectious/inflammatory events ("multiple hits") an inflammatory stress prevails or "inflammatory/pathogen burden" accumulates, which substantially contributes to an enhancement of the inflammatory parameters of natural immune response. Such enhanced inflammatory parameters characterize persons at increased risk of degenerative diseases like atherosclerosis or coronary heart disease. The risk is the higher, the higher the "pathogen burden". An impact of the inflammatory load on cardiac ageing has not yet been described.

"CARDIAC AGEING", REFLECTED BY A NARROWING OF HEART RATE VARIABILITY: The physiological ageing process of the heart goes along with a narrowing of heart rate variability as shown by various groups, including our own. Arguments in favour of a causal relationship between inflammation and cardiac ageing come from an experimental study with healthy human volunteers who had received a low dose of endotoxin: such a proinflammatory stimulus leads to a reversible narrowing of heart rate variability (7). Also in senescence heart rate variability steadily declines, paralleled by a steady increase of basal inflammatory activity.

The reduction of heart rate variability also is regarded as a sensitive parameter of autonomic dysfunction, which contributes to the compromise of cardiac reserve in old age. Apart from typical morphological features and functional deterioration, e.g. diastolic dysfunction, the senescent heart is typically characterized by a narrowed heart rate variability. Efforts have been made to estimate the cardiac age of an individual by this compromised heart rate variability, which may be divergent to the biological age. In recent years diverse approaches were proposed to measure cardiac age on the basis of heart rate variability. The published mathematical formulae were mostly validated with small patient groups and have presently not entered clinical practice. Still heart rate variability is an accepted surrogate parameter of cardiac ageing and is amenable by therapeutic measures, e.g. beta-blockade.

The interaction between autonomic nervous system and inflammation is bilateral: thus vagal stimulation can improve heart rate variability and at the same time evoke anti-inflammatory action: this "cholinergic anti-inflammatory" reflex could make the basis for pharmacological interventions to confine overwhelming inflammatory response syndromes. The afferent vagal nerve, on the other hand, can be stimulated by inflammatory mediators and toxins (endotoxin, Interleukin-1), thus activating the efferent vagus to release acetylcholine, which can bind to a nicotinergic acetylcholine receptor on macrophages and thus interrupt cytokine release and limit the rise in the blood levels of proinflammatory cytokines (TNF, IL-6). The biological meaning of this reflex is to localise inflammatory reactions in the organism and prevent a spill of cytokines to the circulation. A functioning autonomic nervous system is thus mandatory to prevent overshooting of inflammatory response to infection and non-infectious stimuli. The link between cardiac ageing and autonomic dysfunction gives another argument in favour of the notion that autonomic dysfunction and pathogen/inflammatory load could be factors promoting cardiac ageing. This, on the other hand, implies the chance of slowing down the cardiac ageing process by successfully modulating the extent of autonomic dysfunction and the scope of "pathogen/inflammatory burden".

THE NEED FOR A TRIAL:

A possible causal relationship between basal inflammatory activation and cardiac ageing has not been established. This is the issue of the project proposal. In this trial the investigators strive to lower the "pathogen/ inflammatory load" by simple and safe measures. The investigators therefore chose treatment with statins, standardised physical training (both parameters of heart function and heart rate variability could thus be improved) and vaccinations against influenza and pneumococci to prevent a further enhanced "pathogen/ inflammatory burden".

ELIGIBILITY:
Inclusion Criteria:

* age 60-75
* physical activity less than 3 times a week
* written informed consent

Exclusion Criteria:

* heart disease requiring treatment
* treatment with beta-receptor-antagonists
* treatment with statins
* treatment with immunosuppressive drugs
* treatment with anti- inflammatory drugs
* underlying hematological disease
* alcohol abuse, drug abuse
* diabetes mellitus
* study participation within past 30 days
* known intolerance to active agent or any other component of the drug
* active liver disease or unexplained persistent elevation of serum levels of transaminases or cholestasis
* existing myopathy
* pregnancy or nursing period
* absence of an ophthalmological examination within 12 month prior inclusion
* known cataract

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
reduced narrowing of heart rate variability (measured by SDNN of a standardised 20 minute- resting-ecg) via lowering inflammatory/ pathogen burden by anti-inflammatory measures (standardized physical activity and statin administration) | 24 months

SECONDARY OUTCOMES:
quality of life | 24 months
inflammatory parameters | 24 months
major adverse cardiac events (MACE)including death, non lethal myocardial infarction and hospitalisation for cardiovascular reason | 24 month
inflammatory parameters in vaccinated and unvaccinated probands | 24 months
heart rate variability in vaccinated and unvaccinated probands | 24 month
evidence of reduced narrowing of heart rate variability (measured by SDNN of a 24-hours-holter-ecg) via lowering inflammatory/ pathogen burden by anti-inflammatory measures (standardized physical activity and statin administration) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Müller-Werdan, Prof.Dr.med., Study Chair — Martin-Luther-University Halle-Wittenberg, Medical Faculty
Locations (1):
- Martin-Luther-Universität Halle-Wittenberg, Medizinische Fakultät, Klinik und Poliklinik für Innere Medizin III, Universitätsklinikum Halle (Saale), Ernst-Grube-Strasse 40, Halle, Saxony-Anhalt, Germany